CLINICAL TRIAL: NCT02410954
Title: Transcranial Direct Current Stimulation (tDCS) as a Treatment for Acute Fear
Acronym: tDCS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: Pro00059590
Record Dates: First submitted 2015-02-20; First posted 2015-04-08 (Estimated); Results first posted 2021-05-18 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Fear

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No

ARMS (2):
- tDCS electrode configuration (Experimental): Three rounds of tDCS using NeuroConn Direct Current stimulator Multiple Channel -4, Rogue Resolutions treatment optimization where each round includes identifying a promising electrode configuration based on electric field modeling using a realistic head model and capitalizing on the experience with the prior round (for rounds 2 and 3) and testing that electrode placement by administering a series of electrical doses of tDCS with that tDCS electrode configuration (carrying out a dose titration) in a cohort of 10 healthy control subjects to see if we can find an electrical dose which is well-tolerated, safe, suppresses the AOT pupil response and is below recommended current density safety limits (the safety limit in terms of Amperage varies depending on the electrode configuration)
  Interventions: Device: NeuroConn Direct Current stimulator Multiple Channel -4
- Using tDCS to reduce acute fear (Placebo Comparator): Administration of 7.5% CO2 to see if this elicits symptoms of Acute Fear and activates LC and whether tDCS safely inhibits the LC response to 7.5% CO2 compared with sham in a pilot cross-over trial (N=10). A 3-year double-blind, randomized, controlled trial where clinical symptoms of Acute Fear, the primary outcome are elicited with 7.5% CO2 in healthy volunteers is the final study component.
  Interventions: Device: NeuroConn Direct Current stimulator Multiple Channel -4

INTERVENTIONS:
Device: NeuroConn Direct Current stimulator Multiple Channel -4 — (tDCS) will be administered with a multichannel tDCS device that can be programmed so that the operator doesn't know the combination of electrodes being used for stimulation, and, thereby allow double-blinding. The active tDCS electrode configuration to be used will be determined with the 3 round iterative procedure described above; based on electric field modeling and personalized electrical dose titration to find the lowest dose that is well-tolerated and engages the target in terms of inhibiting the AOT pupillary response.

SUMMARY:
Locus coeruleus (LC) norepinephrine (NE) neuron activity has been convincingly linked to regulation of acute fear. This study will address whether LC NE activity examined through pupil measures will reflect carbon dioxide (CO2) induced fear-responses in humans and if transcranial direct current stimulation (tDCS) can mitigate these effects. A 2 year R21 phase establishing feasibility, tolerability, safety, and proof-of-concept (POC) in terms of capacity to engage LC NE neurons with tDCS, followed by a 3 year R33 parallel-group, double-blind, randomized, controlled trial will determine the degree to which engaging LC NE neurons with tDCS improves clinical symptoms.

DETAILED DESCRIPTION:
The National Institutes of Mental Health (NIMH) has recently identified that a major limitation to the understanding of neuropsychiatric disorders and the development of treatments for these conditions has been the inability to identify key dimensions of observable behavior that are central to these disorders and linked to underlying neurobiology by measurable biomarkers. This project is intended to address this problem by establishing that pupillary measures of norepinephrine (NE) neuronal activity are biomarkers of fear dimension of observable behavior, alterations of which are believed to be core features of neuropsychiatric conditions such as anxiety disorders. The investigators will establish this biomarker-clinical dimension link by comparing pupillary indices in humans to a carbon dioxide (CO2) fear provocation test, as well as in these subjects undergoing transcranial Direct Current Stimulation (tDCS) prior to and after CO2 administration.

Participants will be recruited in Dr. Krystal's laboratory at Duke University which has proven infrastructure for clinical trials. The study team plans to enroll a total of 240 subjects healthy volunteers (age range: 21-65 years) in order to complete 100. This takes into account the expected rate of failure to: have a pupillary response in the auditory oddball task (AOT) (25%); have a sufficient fear response to CO2 challenge (50% - relevant for last 10 R21 and all R33 subjects); and to meet other screening criteria.

R21 Phase: First 30 Subjects will undergo two sessions separated by 1 week in which a promising electrode configuration (three promising configuration will each be tested in a cohort of 10 subjects) will be used with tDCS stimulation at increasing electrical dosage during which pupillometry will be carried out to determine the auditory oddball test (AOT) response. A maximum of 5 total tDCS dosages and sham will be tested. Last 10 Subjects. These subjects will take part in a double-blind, controlled, randomized, cross-over study over 3 sessions. At session 1 subjects will undergo electrical dose titration with the tDCS electrode configuration resulting from the 3 rounds of optimization using the same procedure as in the first 30 subjects to determine the lowest well-tolerated dose that suppresses the AOT pupil response, except that a maximum of 5 tDCS dosages will be tested at this session. At the third and fourth sessions (1 week apart) subjects will receive dose-optimized tDCS and the control treatment with order randomized along with 7.5% CO2 (to evoke an LC response) for 20 minutes. The 7.5% CO2 will be delivered to us pre-mixed provided by Airgas. At these sessions, the VAS-A and State Trait Anxiety-Inventory (STA-I) will be administered 5 minutes prior to and just after the 20 minute session and Visual Analog Scale-Anxiety (VAS-A) will also be obtained at 5, 10, 15, and 20 minute points of the CO2 inhalation. tDCS will be administered during the last 5 minutes of the 20 minute CO2 inhalation period. Subjects will be monitored for an hour post-session for safety and will undergo study physician assessment to determine suitability to leave. Following the 2nd treatment session participation will end except that subjects will be called the next day to assess for adverse effects and appropriate care will be given if found. R33 Phase: 60 subjects will participate in a double-blind, randomized, controlled, parallel-group trial. They will be randomized to either active or control treatment and at the first post-screening visit they will undergo electrical dose titration as described above for the treatment they are randomized to. For all titrations, during the 5 minutes between tDCS treatments an unblinded member of the study team not having contact with the subjects will compute their AOT pupil response and convey to the tDCS treatment physician whether to continue or stop titration. Subjects randomized to the control treatment will undergo a sham titration where the stop level will be randomly selected from the distribution of titration outcomes occurring in the R21 phase. Subjects will then return in 1 week and undergo optimal dose tDCS or control treatment for a single treatment session as described in the prior paragraph. Primary outcome will be the VAS-A "fearful" rating obtained at the end of tDCS/CO2 inhalation. AOT pupil response will be obtained every 10 minutes after the end of the tDCS/CO2 inhalation period to map the duration of persistent effects on LC. At the end of this session participation will end except that subjects will be called the next day to assess for adverse effects and care given if necessary. Preliminary data from the R21 phase will be used to provide justification for the larger R33 study, and prior to commencing the R33 investigation phase that an addendum to the Institutional Review Board (IRB) protocol with approval will be obtained.

Pupillometry Procedure. The team will employ fully mobile SensoMotoric Instruments (SMI) Eye-tracking Glasses to carry out pupillometry. Pupil diameter will be recorded continuously from the each eye at a sampling rate of 60 Hz via glasses on the subject's face. The investigators will capture pupil size at baseline and in response to the AOT and administration of 7.5% CO2. Data will be segmented into epochs from 0 to 12 s relative to the acquisition onset of each stimuli or experimental condition. An average pupil diameter measure will then be calculated for the corresponding volume by taking the mean across the remaining non-artifactual samples in that epoch. For 7.5% CO2 response the pupil diameter will be averaged over 1 minute periods while subjects are staring at a dark screen in a dark room. This will be computed at baseline, and at 5, 10, 15, and 20 minutes after the start of CO2 inhalation and 5 minutes and 30 minutes postinhalation.

Administration of 7.5% CO2. Inhalation of 7.5% CO2 for 20 min will be carried out. Subjects will be instructed to avoid alcohol for 36 hours and caffeine for 12 hour prior to testing and to eat a light lunch at least one hour prior to testing. A urine pregnancy test will be administered to women of childbearing potential on both days of gas exposure with a negative result needed in order to continue in study participation. Gas will be delivered via a nasal-oral face mask connected via tubing to a 500 L reservoir bag filled with 7.5% CO2/21% Oxygen (O2) 71.5% Nitrogen (N2). Subjects will receive air through the mask in the 10 min prior to CO2 administration during which baseline measures will be obtained.

Transcranial Direct Current Stimulation (tDCS) will be administered with a multichannel direct current stimulation device that can be programmed so that the operator doesn't know the combination of electrodes being used for stimulation, and, thereby allow double-blinding. The active tDCS electrode configuration to be used will be determined with the 3 round iterative procedure described above; based on electric field modeling and personalized electrical dose titration to find the lowest dose that is well-tolerated and engages the target in terms of inhibiting the AOT pupillary response. Electrical dosage will be personalized for each subject by titrating dosage (gradually increasing) until the dosage is found that is both well-tolerated (no more than mild discomfort on a 5-point Likert scale) and suppresses the AOT pupillary response. If the 5-point Likert tolerability rating is greater than "mild discomfort" or if maximum amperage is reached without effect on AOT then subject participation will terminate.

ELIGIBILITY:
Inclusion Criteria:

* Use of effective method of birth control for women of childbearing capacity
* Willing and able to provide informed consent
* Have a significant difference between the mean pupil diameter in response to odd and common tones in the AOT during screening
* The10 subjects in the R21 cross-over study and all of the R33 subjects must have a 26% increase in VAS-A "fearful" response to 7.5% CO2 at the first CO2 challenge session
* Able to follow study procedures.

Exclusion Criteria:

* Current or past Axis I Diagnostic and Statistical Manual (DSM-IV) disorder based on the MINI
* Current or past history of substance abuse or dependence (excluding nicotine) based on history or positive urine toxicology
* Current unstable medical condition
* Any current neurological condition or medical condition that is known to affect pupillary function, mood/anxiety, or neurologic function generally
* Pregnancy based on Urine Pregnancy Test
* Women who are breast-feeding
* Use of medications known to affect Central Nervous System (CNS) function within 5 half-lives screening
* Use of a pacemaker

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-12; Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Krystal, MD, MS, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Insel TR. The NIMH Research Domain Criteria (RDoC) Project: precision medicine for psychiatry. Am J Psychiatry. 2014 Apr;171(4):395-7. doi: 10.1176/appi.ajp.2014.14020138. No abstract available. PMID 24687194
- [Background] Cuthbert BN, Insel TR. Toward the future of psychiatric diagnosis: the seven pillars of RDoC. BMC Med. 2013 May 14;11:126. doi: 10.1186/1741-7015-11-126. PMID 23672542
- [Background] Redmond DE Jr, Huang YH. Current concepts. II. New evidence for a locus coeruleus-norepinephrine connection with anxiety. Life Sci. 1979 Dec 24;25(26):2149-62. doi: 10.1016/0024-3205(79)90087-0. No abstract available. PMID 120478
- [Background] Nutt DJ. Altered central alpha 2-adrenoceptor sensitivity in panic disorder. Arch Gen Psychiatry. 1989 Feb;46(2):165-9. doi: 10.1001/archpsyc.1989.01810020067011. PMID 2536539
- [Background] LeDoux J. Emotional networks and motor control: a fearful view. Prog Brain Res. 1996;107:437-46. doi: 10.1016/s0079-6123(08)61880-4. No abstract available. PMID 8782535
- [Background] Gilzenrat MS, Nieuwenhuis S, Jepma M, Cohen JD. Pupil diameter tracks changes in control state predicted by the adaptive gain theory of locus coeruleus function. Cogn Affect Behav Neurosci. 2010 May;10(2):252-69. doi: 10.3758/CABN.10.2.252. PMID 20498349
- [Background] Nieuwenhuis S, Aston-Jones G, Cohen JD. Decision making, the P3, and the locus coeruleus-norepinephrine system. Psychol Bull. 2005 Jul;131(4):510-32. doi: 10.1037/0033-2909.131.4.510. PMID 16060800
- [Background] Aston-Jones G, Cohen JD. Adaptive gain and the role of the locus coeruleus-norepinephrine system in optimal performance. J Comp Neurol. 2005 Dec 5;493(1):99-110. doi: 10.1002/cne.20723. PMID 16254995
- [Background] Bailey JE, Argyropoulos SV, Kendrick AH, Nutt DJ. Behavioral and cardiovascular effects of 7.5% CO2 in human volunteers. Depress Anxiety. 2005;21(1):18-25. doi: 10.1002/da.20048. PMID 15782425
- [Background] Biancardi V, Bicego KC, Almeida MC, Gargaglioni LH. Locus coeruleus noradrenergic neurons and CO2 drive to breathing. Pflugers Arch. 2008 Mar;455(6):1119-28. doi: 10.1007/s00424-007-0338-8. Epub 2007 Sep 13. PMID 17851683
- [Background] Pineda J, Aghajanian GK. Carbon dioxide regulates the tonic activity of locus coeruleus neurons by modulating a proton- and polyamine-sensitive inward rectifier potassium current. Neuroscience. 1997 Apr;77(3):723-43. doi: 10.1016/s0306-4522(96)00485-x. PMID 9070748

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | tDCS Electrode Configuration | Using tDCS to Reduce Acute Fear
Started | 14 | 0
Completed | 0 | 0
Not Completed | 14 | 0
Not completed — Unable to collect usable data due to initial protocol issues | 6 | 0
Not completed — Instrument malfunction generated unusable data | 8 | 0

BASELINE CHARACTERISTICS:
Population: The tDCS electrode configuration study was terminated prematurely due to technical problems and delay due to a move. The Using tDCS to reduce acute fear study was never started as a result.
Groups:
- Total: Total of all reporting groups
Arm/Group | tDCS Electrode Configuration | Using tDCS to Reduce Acute Fear | Total
Number analyzed (Participants) | 14 | 0 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 14 |  | 14
  >=65 years | 0 |  | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 |  | 9
  Male | 5 |  | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 9 | 0 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 |  | 14

OUTCOME MEASURES:

1. Primary Outcome: Change in VAS-A Rating
Description: Primary outcome will be the VAS-A "fearful" rating obtained at the end of tDCS/CO2 inhalation. AOT pupil response will be obtained every 10 minutes after the end of the tDCS/CO2 inhalation period to map the duration of persistent effects on LC.
Time Frame: Every 10 min (for approximately 20 minutes) at the end of tDCS/CO2 inhalation following one week post stimulation optimization.
Population: No data are available to report as the instrument used malfunctioned and did not produce usable pupil measurements.
Arm/Group | tDCS Electrode Configuration | Using tDCS to Reduce Acute Fear
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 month
Description: No differences
Arm/Group | tDCS Electrode Configuration | Using tDCS to Reduce Acute Fear
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/0
Other Adverse Events (participants affected / at risk) | 0/14 | 0/0

LIMITATIONS AND CAVEATS:
Study terminated prematurely without generating any outcome data due to delays due to the study being moved from one institution to another and due to technical problems with the pupil measurements that required a long period of trouble-shooting/problem-solving and ultimately the replacement of the pupillometry device.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-06): https://cdn.clinicaltrials.gov/large-docs/54/NCT02410954/Prot_SAP_000.pdf